CLINICAL TRIAL: NCT06807710
Title: A Study on the Effects of Dynamic Neuromuscular Stabilization Exercises on Pain, Posture, and Respiratory Muscle Strength in Individuals With Chronic Non-Specific Low Back Pain
Brief Title: Effects of Dynamic Neuromuscular Stabilization on Pain, Posture, and Respiratory Strength in Chronic Low Back Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, MERVE BAŞARDI, Physiotherapist, Uskudar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-PT-MRVB-RCT
Record Dates: First submitted 2025-01-29; First posted 2025-02-04 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Chronic Low-back Pain
Keywords: Rehabilitation; Exercise Therapy; Physiotherapy

STUDY DESIGN:
Intervention Model Description: Training and Control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DNS Group (Experimental): Participants diagnosed with chronic non-specific low back pain will undergo a structured dynamic neuromuscular stabilization (DNS) exercise program. The intervention will be conducted twice a week, with each session lasting 45 minutes, over a period of 8 weeks. The program will focus on improving motor control, spinal stability, and neuromuscular coordination through DNS principles.
  Interventions: Other: DNS Group
- Pilates Group (Experimental): Participants in this group will perform Reformer Pilates exercises designed to improve core stability, flexibility, and overall postural alignment. The intervention will also be conducted twice a week, with each session lasting 45 minutes, over a period of 8 weeks. Exercises will target strengthening the deep stabilizing muscles and enhancing spinal mobility while maintaining a controlled and safe environment.
  Interventions: Other: Pilates Group

INTERVENTIONS:
Other: DNS Group — Dynamic neuromuscular stabilization exercises, on the other hand, are designed to achieve sagittal stabilization by utilizing the stabilizing function of the thoracic diaphragm muscle.
  Other Names: Dynamic Neuromuscular Stabilization
  Arms: DNS Group
Other: Pilates Group — Reformer pilates exercises, focusing on core stability, flexibility, postural alignment, and breath control using a Reformer Pilates machine under the supervision of a physiotherapist.
  Other Names: Reformer Pilates Exercise
  Arms: Pilates Group

SUMMARY:
This study aims to evaluate the effects of dynamic neuromuscular stabilization exercises on individuals experiencing chronic non-specific low back pain for at least six months. Pain intensity will be assessed using the Visual Analog Scale (VAS) marked on a 10 centimeter line. The impact of low back pain on daily activities will be evaluated through the Oswestry Disability Index, while its influence on quality of life will be determined using the Short Form-36 (SF-36). Postural changes related to low back pain will be assessed using the New York Posture Scale. The effects on respiratory muscles will be examined through lung volume measurements using a spirometer, and respiratory patterns will be identified using chest circumference measurements with a measuring tape.

DETAILED DESCRIPTION:
This study investigates the effects of dynamic neuromuscular stabilization (DNS) exercises on pain, posture, and respiratory muscle strength in individuals with chronic non-specific low back pain. Participants with low back pain persisting for at least six months will be included in the study. The primary objective is to assess the impact of DNS exercises on pain intensity, functional disability, quality of life, posture, and respiratory function.

Pain intensity will be measured using the Visual Analog Scale (VAS) on a 10-centimeter line. Functional disability related to low back pain will be evaluated using the Oswestry Disability Index, a reliable and valid tool for assessing the impact of back pain on daily activities. Quality of life will be measured using the Short Form-36 (SF-36), a comprehensive instrument assessing physical and mental health dimensions.

To evaluate postural changes, the New York Posture Scale will be employed, providing a systematic approach to assess spinal alignment and postural deviations. The study will also examine the effects of DNS exercises on respiratory muscle performance and lung function. Lung volumes will be measured using a spirometer, while respiratory patterns will be analyzed by chest circumference measurements at different thoracic levels using a measuring tape.

The intervention will involve a structured exercise program based on DNS principles, focusing on improving motor control, spinal stability, and neuromuscular coordination. Participants will be assessed at baseline and post-intervention, with follow-up evaluations conducted to observe the long-term effects of the intervention. The study aims to contribute to the understanding of DNS as an effective approach for managing chronic non-specific low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 50 years
* Experiencing continuous or intermittent low back pain for more than 3 months, localized between the L1 region and gluteal muscles

Exclusion Criteria:

* Specific medical diagnoses such as spinal fractures or spinal stenosis
* Presence of rheumatological disorders
* Tumors
* History of lumbar surgery in the last 3 years
* Neurological problems
* Osteoporosis
* History of epilepsy, vertigo, headaches, or nausea
* Chronic lung diseases
* Prior physiotherapy treatment for low back pain
* Acute low back pain episodes
* Mental disorders
* Pregnancy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-03 (Estimated); Primary Completion 2025-05-03 (Estimated); Study Completion 2025-07-03 (Estimated)

PRIMARY OUTCOMES:
Respiratory Muscle Strength | 8 weeks
  Respiratory muscle strength was measured using an electronic mouth pressure measuring device (Cosmed Ponyy Fx, Rome, Italy). Maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP) were measured.
Visual Analog Scale (VAS) | 8 weeks
  The Visual Analog Scale (VAS) will be used to measure pain intensity by having participants mark their perceived level of pain on a 10-centimeter line ranging from 'no pain' to 'worst pain imaginable. The Visual Analog Scale (VAS) for pain ranges from a minimum of 0 to a maximum of 10, with higher scores indicating greater pain intensity.
New York Posture Analysis | 8 weeks
  The New York Posture Analysis is a validated and systematic tool used to evaluate postural alignment and deviations. This method involves visual inspection and scoring of key postural elements, including head, shoulders, spine, pelvis, and lower extremities, in both anterior-posterior and lateral views. Each segment is assessed for alignment and assigned a score based on observed deviations. The total score reflects the overall postural status, with higher scores indicating better postural alignment. This measure will be used to assess changes in posture pre- and post-intervention. The New York Posture Rating Scale scores range from a minimum of 0 to a maximum of 36, with higher scores indicating better posture.

SECONDARY OUTCOMES:
Oswestry Disability Index (ODI) | 8 weeks
  he Oswestry Disability Index is a self-reported questionnaire designed to assess how low back pain affects an individual's ability to perform daily activities. The index consists of 10 sections, each addressing a specific domain: pain intensity, personal care, lifting, walking, sitting, standing, sleeping, sexual life, traveling, and social life. Each section includes six response options scored from 0 (no disability) to 5 (maximum disability). The total score ranges from 0 to 50 points, with higher scores indicating greater levels of disability.
Short Form-36 (SF-36) Health Survey | 8 weeks
  The Short Form-36 (SF-36) Health Survey is a widely used self-reported questionnaire designed to assess health-related quality of life across eight domains: physical functioning, role limitations due to physical health, role limitations due to emotional health, energy/fatigue, emotional well-being, social functioning, pain, and general health perceptions. Each domain is scored on a scale from 0 to 100, with higher scores indicating better health and quality of life.
Chest Circumference Measurement | 8 weeks
  Chest circumference measurement is a simple and reliable method used to assess respiratory patterns and chest expansion. Measurements will be taken at three levels: axillary (upper thoracic), xiphoid (middle thoracic), and subcostal (lower thoracic) regions using a measuring tape. The difference between maximum inspiration and maximum expiration at each level will be recorded to determine the chest expansion.

CONTACTS AND LOCATIONS:
Overall Officials: Filiz Eyuboglu, PhD., Study Director — Uskudar University; Mert Ilhan, MSc., Principal Investigator — Uskudar University
Locations (1):
- Uskudar University Physiotherapy and Rehabilitation Application and Research Center, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No